CLINICAL TRIAL: NCT06666348
Title: A Phase 1/2 Study of Mirdametinib and Vinblastine for Newly Diagnosed or Previously Untreated Patients With Pediatric Low-grade Glioma and Activation of the MAPK Pathway
Brief Title: Phase 1/2 Study of Mirdametinib + Vinblastine for Newly Diagnosed/Previously Untreated PLGG + Activation of MAPK
Acronym: MIRV
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Dr Perreault, Principal Investigator, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRV
Record Dates: First submitted 2024-10-09; First posted 2024-10-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Low-grade Glioma
Keywords: PLGG; Pediatric PLGG; Pediatric; MAPK; NF1; KIAA1549-BRAF; pediatric low-grade glioma
MeSH Terms: interventions — mirdametinib; Vinblastine

STUDY DESIGN:
Intervention Model Description: This is a 3-part open-label study (feasibility phase, treatment phase and follow-up phase) of orally administered mirdametinib in combination with intravenous vinblastine chemotherapy in patients with PLGG with activation of MAPK pathway.
  Feasibility Phase:
  The maximum tolerated/recommended phase 2 dose (MTD/RP2D) of the mirdametinib plus vinblastine combination will be assessed using a modified Rolling-6 design.
  Treatment Phase:
  Patients will receive mirdametinib twice daily (continuously) at a fixed dose (2mg/m2 po BID up to 4 mg BID) for a total of 13 cycles (28 days cycle). Weekly intravenous vinblastine at MTD will be given for a total of 17 cycles. If adverse events occur, two dose reductions are allowed.
  Follow-up Phase:
  Following the end of treatment, patients will be scheduled for a follow-up visit every 6 months for 36 months to evaluate PFS, TTP and OS.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Mirdametinib + IV Vinblastine (Experimental): Patients will receive oral mirdametinib twice daily (continuous) at a fixed dose (2mg/m2 PO BID, rounded to the nearest 1mg, up to a maximum of 4 mg BID) for a total of 13 cycles. Each cycle will last 28 days.
  Interventions: Drug: Mirdametinib

INTERVENTIONS:
Drug: Mirdametinib — Participants will receive orally administered mirdametinib in combination with intravenous vinblastine chemotherapy
  Other Names: Vinblastine

SUMMARY:
This is a 3-part open-label study (feasibility phase, treatment phase and follow-up phase) of orally administered mirdametinib in combination with intravenous vinblastine chemotherapy in patients with PLGG with activation of MAPK pathway.

Feasibility Phase:

The maximum tolerated/recommended phase 2 dose (MTD/RP2D) of the mirdametinib plus vinblastine combination will be assessed using a modified Rolling-6 design.

Treatment Phase:

Patients will receive mirdametinib twice daily (continuously) at a fixed dose (2mg/m2 po BID up to 4 mg BID) for a total of 13 cycles (28 days cycle). Weekly intravenous vinblastine at MTD will be given for a total of 17 cycles. If adverse events occur, two dose reductions are allowed.

Follow-up Phase:

Following the end of treatment, patients will be scheduled for a follow-up visit every 6 months for 36 months to evaluate PFS, TTP and OS.

DETAILED DESCRIPTION:
This is a phase 1/2, open label, interventional clinical trial that will study the response rate of newly diagnosed pediatric low-grade glioma (PLGG) to oral administration of mirdametinib in combination with weekly vinblastine. Patients meeting all inclusion criteria for a given study group will receive mirdametinib twice daily (continuous) at a fixed dose (2 mg/m2 po BID up to 4 mg BID) for a total of 13 cycles (28 days cycle). Weekly intravenous vinblastine at MTD will be given for a total of 17 cycles.

The lead-in feasibility phase will be conducted to establish the maximum tolerated/recommended phase 2 dose (MTD/RP2D) of vinblastine in combination with mirdametinib combination using a modified Rolling-6 design. The established RP2D for mirdametinib (2 mg/m2 po BID up to 4 mg BID) will be used on this study. Mirdametinib will be administered on a continuous dosing schedule and de-escalated as necessary to an intermittent (3 weeks on, 1 week off) dosing schedule. Vinblastine will be escalated (or de-escalated) as necessary. Since these classes of agents do not have overlapping toxicities, the starting dose (i.e., Dose Level 0) for vinblastine is 4 mg/m2/week, which is 20% lower than the recommended single agent dose of vinblastine of 5 mg/m2/week. Dose Level 1 for vinblastine is 5 mg/m2/week and Dose Level -1 for vinblastine is 3 mg/m2/week.

Following the end of treatment, patients will be scheduled for a follow-up visit every 6 months for 36 months to evaluate PFS, TTP and OS. A total of 50 patients will be recruited as part of this clinical study.

Patients aged between 2 and 25 years old will be eligible, in order to include a maximum of patients affected by glioma. This study includes PLGG patients with neurofibromatosis type 1 (NF1) with a KIAA1549-BRAF fusion and patients with activation of the MAPK pathway with the exception of patients with a BRAFV600E mutation.

Response to treatment will be evaluated using the modified Response Assessment in Pediatric Neuro-Oncology (RAPNO), Response Assessment in Pediatric Neuro-Oncology (RANO) 1. Evaluation of quality of life will be measured using the Pediatric Quality of Life inventory (PedsQL) (Generic/Brain tumor modules).

This study will explore the genetic and epigenetic landscape of PLGG. Our biological study may include SNP array, nanoString studies, methylation array and RNAseq.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent prior to study participation.
* Study activities compliance: must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study, including disease assessment by contrast enhanced MRI.
* Aged ≥ 2 years to ≤ 25 years when starting mirdametinib.
* BSA ≥ 0,40m2
* Diagnosis:

Participants must have PLGG with NF1 gene mutation (based on clinical NIH criteria, germline NF1 mutation or molecular analysis of the tumor) or PLGG with KIAA1549-BRAF fusion (based on molecular analysis of the tumor) or PLGG with evidence of MAPK pathway alteration with the exception of patients with BRAF V600E mutation (based on molecular analysis of the tumor).

* Tumor tissue is required (at minimum, paraffin-embedded tissue block and additionally fresh frozen tissue [if available]). Patients with NF1 and Low Grade Glioma (LGG) can still be enrolled without tissue if no surgery or biopsy was conducted.
* Baseline MRI.
* Life expectancy greater than 6 months.
* Lansky/Karnofsky score ≥ 50.
* Normal organ and marrow function (see study protocol for specifics).
* Female and male patients of fertile age must agree to use highly effective contraceptive measures.
* Must be able to ingest by mouth and retain entirely the administered medication. Mirdametinib can not be administered via nasogastric tube or gastrostomy tube.

Exclusion Criteria:

* Patients who are receiving other investigational agents.
* Cardiac: QTcB ≥ 480 msec or an absolute resting left ventricular ejection fraction (LVEF) of ≤ 49%.
* Patients who have any other malignancy, except if the other primary malignancy is neither currently clinically significant nor requiring active intervention.
* Tumor with BRAF V600E mutation.
* Patients who received previous systemic or radiotherapy treatment.
* Other severe and uncontrollable medical disease
* Blood pressure higher than 95th percentile for patient's age, height and gender.
* Increased risk of serious retinopathy and retinal vein occlusion.
* Known diagnosis of human immunodeficiency virus infection, hepatitis B or C.
* Previous major surgery within 2 weeks.
* History of allergic reactions to compounds of similar chemical or biological composition to mirdametinib.
* Pregnant or breastfeeding.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2030-04 (Estimated); Study Completion 2033-04 (Estimated)

PRIMARY OUTCOMES:
Determine maximum tolerated dose of Mirdametinib plus Vinblastine. | 3 years
  The maximum tolerated/recommended phase 2 dose (MTD/RP2D) of the mirdametinib plus vinblastine combination using a modified Rolling-6 design.
Determine the objective response rate of mirdametinib plus vinblastine for PLGG with Mitogen-activated Protein Kinase (MAPK) pathway activation in treatment naïve patients. | 5 years
  The proportion of patients with complete (CR), major (MaR), partial (PR) and minor response (MiR) as the best response on study based on RAPNO criteria.
  Response = MiR+PR+MaR+CR

SECONDARY OUTCOMES:
Efficacy outcome measures: Overall Survival. | Up to 3 years following completion of treatment.
  Overall Survival (OS) is defined as the time from starting mirdametinib (C1D1) to death due to any cause, or censored at date last known alive. OS will be evaluated from starting mirdametinib up to the end of the 3-year follow-up. Estimated using Kaplan-Meier methods.
Efficacy outcome measures: Progression-Free Survival. | Up to 3 years following completion of treatment.
  Progression-Free Survival (PFS): the time from starting mirdametinib (C1D1) to the date of first observation of radiological progression or death due to any cause. Participants alive without disease progression or death are censored at date of last disease evaluation. Estimated using Kaplan-Meier methods.
Efficacy outcome measures: Time to Progression. | Up to 3 years following completion of treatment.
  Time to Progression (TTP) is defined as the time from starting mirdametinib (C1D1) to radiological progression, or censored at date of last disease evaluation for those without progression reported. Estimated using Kaplan-Meier methods.
Efficacy outcome measures: Objective Response Rate. | Up to 3 years following completion of treatment.
  Objective response rate (ORR) is defined as the percentage of patients experiencing their best response on study as CR or PR or MR or SD.
Determine the safety and tolerability of the combination of mirdametinib plus vinblastine. | 5 years
  Adverse events (AE) and severe adverse events (SAE).
Determine neurological changes in patients during active treatment and after completion of therapy. | 5 years
  Changes in neurological status will be evaluated. Standardized global assessment including motor function will be evaluated by local investigators at baseline, every six months during treatment phase and after completion of treatment. This evaluation will include assessment of weakness, coordination, and balance.
Evaluate the quality of life during treatment. | 5 years
  Evaluations of quality of daily life at inclusion and every six months PedsQL (Generic/Brain tumor modules).

OTHER OUTCOMES:
Evaluate the response rate based on the tumor volume. | 5 years
  Accurate quantification of tumor volumes using a semi-automated volumetric method.
To investigate and correlate biological features to tumor response. | 5 years
  Exploratory biology studies may include, but are not limited to: tumor molecular profiling, gene expression, methylation profiling and DNA sequencing to explore possible associations between candidate molecular predictors and clinical outcome.
  Descriptive statistics may be used to visualize biological feature results and compare to measures of efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Perreault, M.D, FRCPC, Study Chair — CHU Sainte Justine, URCHOI Department
Locations (4):
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Childrens and Womens Health Centre of British Columbia - British Columbia Childrens Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Data will be share with researchers upon request following publication of data analysis of trial via scientific articles.
Supporting Information: CSR
Time Frame: 2030-2040
Access Criteria: Upon request to the sponsor and study chair

REFERENCES:
- [Result] Robinson GW, Vinitsky A, Bag AK, et al. LGG-53. RESULTS FROM THE PHASE 1 AND PHASE 1 EXPANSION COHORTS OF SJ901: A PHASE 1/2 TRIAL OF SINGLE-AGENT MIRDAMETINIB (PD-0325901) IN CHILDREN, ADOLESCENTS, AND YOUNG ADULTS WITH LOW-GRADE GLIOMA. Neuro Oncol. 2024; 26(Suppl 4):0
- [Result] Gross AM MC, Warren KE, Widemann BC. Plasma and cerebrospinal fluid pharmacokinetics of selumetinib in non-human primates (NHP). Journal of Clinical Oncology. 2017; 35((15_suppl)):e14070-e14070
- [Result] Lassaletta A, Scheinemann K, Zelcer SM, Hukin J, Wilson BA, Jabado N, Carret AS, Lafay-Cousin L, Larouche V, Hawkins CE, Pond GR, Poskitt K, Keene D, Johnston DL, Eisenstat DD, Krishnatry R, Mistry M, Arnoldo A, Ramaswamy V, Huang A, Bartels U, Tabori U, Bouffet E. Phase II Weekly Vinblastine for Chemotherapy-Naive Children With Progressive Low-Grade Glioma: A Canadian Pediatric Brain Tumor Consortium Study. J Clin Oncol. 2016 Oct 10;34(29):3537-3543. doi: 10.1200/JCO.2016.68.1585. PMID 27573663
- [Result] Fangusaro J, Onar-Thomas A, Young Poussaint T, Lensing S, Ligon AH, Lindeman N, Banerjee A, Kilburn LB, Lenzen A, Pillay-Smiley N, Pollack IF, Robison NJ, Partap S, Qaddoumi I, Landi D, Jones DTW, Stewart CF, Fouladi M, Dunkel IJ. A phase 2 PBTC study of selumetinib for recurrent/progressive pediatric low-grade glioma: Strata 2, 5, and 6 with long-term outcomes on strata 1, 3, and 4. Neuro Oncol. 2025 Oct 14;27(9):2415-2428. doi: 10.1093/neuonc/noaf065. PMID 40241281
- [Result] Fangusaro J, Onar-Thomas A, Young Poussaint T, Wu S, Ligon AH, Lindeman N, Banerjee A, Packer RJ, Kilburn LB, Goldman S, Pollack IF, Qaddoumi I, Jakacki RI, Fisher PG, Dhall G, Baxter P, Kreissman SG, Stewart CF, Jones DTW, Pfister SM, Vezina G, Stern JS, Panigrahy A, Patay Z, Tamrazi B, Jones JY, Haque SS, Enterline DS, Cha S, Fisher MJ, Doyle LA, Smith M, Dunkel IJ, Fouladi M. Selumetinib in paediatric patients with BRAF-aberrant or neurofibromatosis type 1-associated recurrent, refractory, or progressive low-grade glioma: a multicentre, phase 2 trial. Lancet Oncol. 2019 Jul;20(7):1011-1022. doi: 10.1016/S1470-2045(19)30277-3. Epub 2019 May 28. PMID 31151904
- [Result] Weiss BD, Wolters PL, Plotkin SR, Widemann BC, Tonsgard JH, Blakeley J, Allen JC, Schorry E, Korf B, Robison NJ, Goldman S, Vinks AA, Emoto C, Fukuda T, Robinson CT, Cutter G, Edwards L, Dombi E, Ratner N, Packer R, Fisher MJ. NF106: A Neurofibromatosis Clinical Trials Consortium Phase II Trial of the MEK Inhibitor Mirdametinib (PD-0325901) in Adolescents and Adults With NF1-Related Plexiform Neurofibromas. J Clin Oncol. 2021 Mar 1;39(7):797-806. doi: 10.1200/JCO.20.02220. Epub 2021 Jan 28. PMID 33507822
- [Result] Jones DT, Gronych J, Lichter P, Witt O, Pfister SM. MAPK pathway activation in pilocytic astrocytoma. Cell Mol Life Sci. 2012 Jun;69(11):1799-811. doi: 10.1007/s00018-011-0898-9. Epub 2011 Dec 13. PMID 22159586
- [Result] Packer RJ, Lange B, Ater J, Nicholson HS, Allen J, Walker R, Prados M, Jakacki R, Reaman G, Needles MN, et al. Carboplatin and vincristine for recurrent and newly diagnosed low-grade gliomas of childhood. J Clin Oncol. 1993 May;11(5):850-6. doi: 10.1200/JCO.1993.11.5.850. PMID 8487049
- [Result] Sievert AJ, Fisher MJ. Pediatric low-grade gliomas. J Child Neurol. 2009 Nov;24(11):1397-408. doi: 10.1177/0883073809342005. PMID 19841428
- [Result] Fangusaro J, Witt O, Hernaiz Driever P, Bag AK, de Blank P, Kadom N, Kilburn L, Lober RM, Robison NJ, Fisher MJ, Packer RJ, Young Poussaint T, Papusha L, Avula S, Brandes AA, Bouffet E, Bowers D, Artemov A, Chintagumpala M, Zurakowski D, van den Bent M, Bison B, Yeom KW, Taal W, Warren KE. Response assessment in paediatric low-grade glioma: recommendations from the Response Assessment in Pediatric Neuro-Oncology (RAPNO) working group. Lancet Oncol. 2020 Jun;21(6):e305-e316. doi: 10.1016/S1470-2045(20)30064-4. PMID 32502457